CLINICAL TRIAL: NCT01635036
Title: Eeva 12-well Dish Study
Acronym: NDS
Status: Completed | Type: Observational
Sponsor: Progyny, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2012-AUX-001; TST-1736-p (Other: Auxogyn, Inc.)
Record Dates: First submitted 2012-07-02; First posted 2012-07-06 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Infertility
Keywords: in vitro fertilization; assisted reproduction techniques; noninvasive imaging of embryos; time lapse imaging of embryos; traditional morphological grading of embryos; prediction of blastocyst formation; infertility; male factor female factor; embryo viability
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women undergoing IVF treatment: Women undergoing IVF treatment
  Interventions: Device: In-vitro fertilization using Eeva

INTERVENTIONS:
Device: In-vitro fertilization using Eeva — Eeva will image embryos through cleavage stage (Day 3). Embryologists will use Eeva results along with traditional morphological grading to assist in selecting embryo(s) for transfer or freezing.

SUMMARY:
The purpose of this study is to demonstrate that the Eeva™ System is compatible with the Eeva 12-well Dish.

DETAILED DESCRIPTION:
This study is designed to demonstrate that the Eeva System Software successfully tracks the embryo images and identifies the timing of key developmental events using the Eeva 12-well Dish.

This is a prospective, observational, blinded, single arm, nonrandomized, single center clinical study. Images of developing embryos and Eeva predictions will be blinded to embryologists and physicians

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing fresh in vitro fertilization treatment using their own eggs or donor eggs.
* Subject is at least 18 years of age.
* Subject has basal antral follicle count (BAFC) ≥ 12 prior to stimulation cycle.
* Subjects has basal FSH < 11 IU
* Fertilization using only ejaculated sperm (fresh or frozen) - no surgically removed sperm.
* Subject has at least 8 normally fertilized eggs (2PN)
* Willing to have all 2PN embryos monitored by Eeva
* Willing to comply with study protocol and procedures and able to speak English.
* Willing to provide written informed consent.

Exclusion Criteria:

* Reinseminated eggs.
* History of cancer.
* Gestational carriers.
* Planned preimplantation genetic diagnosis or preimplantation genetic screening.
* Previously enrolled in this study
* Concurrent participation in another clinical study.
* Any other reason the Investigator believes the subject should not participate in the clinical study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women in the United States who undergo IVF treatment
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
To validate and develop the Eeva Software. | 3 months
  The clinical image data (embryos images) will be used to develop the Eeva System Software. The Eeva software validation will consist in comparing the specificity of the Eeva System Software Blastocyst Prediction from the Eeva 12-well Dish to the specificity of the Eeva System Software from the Eeva 25-well Dish (the specificity of the Eeva System Software from the Eeva 25-well Dish was previously determined during the Eeva System Study TST-1788-r).

SECONDARY OUTCOMES:
Specificity and sensitivity and 95% confidence intervals of the Eeva System Software and the Embryologist Panel (also referred to as Panel) measurements will be computed. | 3 months

OTHER OUTCOMES:
The postive/negative (in-window/out-window) agreement of the Eeva Software and Panel measurements will be compared. | 3 months
The Mean Absolute Difference (MAD) will be calculated between each observer (Eeva Software, Panelist 1, Panelist 2, and Panelist 3) | 3 months
Bland Altman plots for the differences between each observer. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Boostanfar, MD, Principal Investigator — HRC Fertility
Locations (1):
- HRC Fertility, Encino, California, United States